CLINICAL TRIAL: NCT07148960
Title: Does Staphylococcus Aureus Bacteremia Early Dual Therapy Improve Outcomes? (SABEDTIO) Clinical Trial
Brief Title: Does Staphylococcus Aureus Bacteremia Early Dual Therapy Improve Outcomes?
Acronym: SABEDTIO
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Joy J. Juskowich, MD, Assistant Professor and COpAT Medical Director, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2507187207
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: MRSA; MSSA
MeSH Terms: interventions — Daptomycin; Ceftaroline; Rifampin; Cefazolin; Ertapenem; Vancomycin; Oxacillin; Nafcillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Dual IV Antibiotic Therapy (Experimental): Once type of Staphylococcus aureus bacteremia (MRSA vs. MSSA) is determined the following IV antibiotics will be given:
  * MRSA - daptomycin plus ceftaroline;
  * MSSA - cefazolin plus ertapenem;
  * MRSA or MSSA - rifampin PO may be added for patients with prosthetic material
  Interventions: Drug: Early Dual IV Antibiotic Therapy - MRSA; Drug: Early Dual IV Antibiotic Therapy - MSSA
- Single Agent IV Antibiotic Therapy (Active Comparator): Once type of Staphylococcus aureus bacteremia (MRSA vs. MSSA) is determined the following IV antibiotics will be given:
  * MRSA - daptomycin, vancomycin, or ceftaroline;
  * MSSA - cefazolin, oxacillin, or nafcillin;
  * MRSA or MSSA - rifampin PO may be added for patients with prosthetic material
  Interventions: Drug: Single Agent IV Antibiotic Therapy - MRSA; Drug: Single Agent IV Antibiotic Therapy - MSSA

INTERVENTIONS:
Drug: Early Dual IV Antibiotic Therapy - MRSA — Participant given IV daptomycin plus ceftaroline dosing per standard of care. Oral rifampin may be added for participants with prosthetic material.
  Other Names: daptomycin; ceftaroline; rifampin
  Arms: Early Dual IV Antibiotic Therapy
Drug: Early Dual IV Antibiotic Therapy - MSSA — Participant given IV cefazolin plus ertapenem dosing per standard of care. Oral rifampin may be added for participants with prosthetic material.
  Other Names: cefazolin; ertapenem; rifampin
  Arms: Early Dual IV Antibiotic Therapy
Drug: Single Agent IV Antibiotic Therapy - MRSA — Participant given one of the following IV therapies: daptomycin, vancomycin, or ceftaroline. Oral rifampin may be added for participants with prosthetic material.
  Other Names: daptomycin; vancomycin; ceftaroline; rifampin
  Arms: Single Agent IV Antibiotic Therapy
Drug: Single Agent IV Antibiotic Therapy - MSSA — Participant given one of the following IV therapies: cefazolin, oxacillin, or nafcillin. Oral rifampin may be added for participants with prosthetic material.
  Other Names: cefazolin; oxacillin; nafcillin; rifampin
  Arms: Single Agent IV Antibiotic Therapy

SUMMARY:
The goal of this open-label, pragmatic, randomized controlled clinical trial is to learn if patients with Staphylococcus aureus bacteremia (SAB) given the intervention of early dual intravenous (IV) antibiotic therapy will decrease duration of bacteremia (< 6 days) and improve outcomes compared to single IV antibiotic therapy.

The main questions this study aims to answer are:

* To decrease SAB duration and improve outcomes by using early dual vs. single agent IV antibiotic therapy
* To accelerate practice transformation of earlier IV to oral (PO) antibiotic transition by switching to PO antibiotic therapy once blood cultures are negative at 72 hours

Participants will be asked to agree to be randomized (like flipping a coin) to receive two or one IV antibiotic(s). Once the infection has cleared, the treatment will be changed to PO antibiotics. As part of usual care, participants will have weekly lab tests for monitoring while on antibiotics, receive a telephone call to see how the participants are doing, and follow up in person or by telephone or video in Infectious Diseases (ID) Clinic. Participant participation will last 12 weeks after the participant is discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* The patient is hospitalized at J.W. Ruby Memorial Hospital, Berkeley Medical Center, Camden Clark Medical Center, Princeton Community Hospital, Thomas Hospital, United Hospital Center, or Wheeling Hospital
* The patient has been identified to have Staphylococcus aureus bacteremia
* The patient is able to participate in lab monitoring and in-person or telemedicine ID Clinic follow-up

Exclusion Criteria:

* The patient or an appointed medical decision maker is unable to give informed consent
* The patient is a prisoner, pregnant, and/or mentally handicapped
* The patient is determined unsafe for enrollment at the primary team's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with prolonged bacteremia (≥ 6 days) | Up to 12 weeks post hospital discharge
  Percentage of participants with prolonged bacteremia (≥ 6 days) up to 12 weeks post hospital discharge.
Seeding of a New Site - Incidence | Up to 12 weeks post hospital discharge
  Incidence of new infection of heart valve, joint, or spine up to 12 weeks post hospital discharge.
All-Cause Mortality | Up to 12 weeks post hospital discharge
  Number of participants who died from any cause up to 12 weeks post hospital discharge.

SECONDARY OUTCOMES:
Number of patients with cure/control | Up to 12 weeks post hospital discharge
  Number of patients with cure/control using clinical (resolution of infection - e.g., wound healed) and laboratory (improvement in inflammatory markers - e.g., CRP normalization) parameters.
Time to Positivity (TTP) | Up to 14 days post hospital admission
  Time in hours from first set of blood culture bottle on laboratory instrument to positive culture bottle off laboratory instrument (TTP1).
Sequential Time to Positivity (STTP) | Up to 14 days post hospital admission
  Ratio of the Time to Positivity of the second set of blood cultures divided by the first set of blood cultures (TTP2/TTP1).
Length of Hospital Stay | Up to 12 weeks post hospital discharge
  Duration in days from hospital admission to hospital discharge.
Overall Hospital Readmission | Up to 12 weeks post hospital discharge
  Number of participants readmitted for any reason up to 12 weeks after discharge from the hospital.
Rate of Relapsed Bacteremia | Up to 12 weeks post hospital discharge
  Recurrence of bacteremia with the same organism one week after initial clearance.
Time to First Negative Blood Culture | Up to 14 days post hospital admission
  Time from hospital admission to the first documented negative blood culture.
Incidence of Antibiotic-Associated Side Effects and Toxicity | Up to 12 weeks post hospital discharge
  Occurrence of adverse events related to antibiotic therapy, including Clostridioides difficile infection, as assessed by clinical evaluation and laboratory testing.

CONTACTS AND LOCATIONS:
Overall Officials: Joy J Juskowich, MD, Principal Investigator — West Virginia University; Arif R Sawari, MD, MSc, MBA, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim M, Ranganath N, Chesdachai S, Stevens RW, Sohail MR, Abu Saleh OM. Which trial do we need? Combination therapy with daptomycin plus ceftaroline versus standard-of-care monotherapy in the treatment of methicillin-resistant Staphylococcus aureus bacteraemia. Clin Microbiol Infect. 2025 Jan;31(1):18-21. doi: 10.1016/j.cmi.2024.08.011. Epub 2024 Sep 7. No abstract available. PMID 39182576
- [Background] Juskowich JJ, Thompson JM, Bage SD, Palmateer KM, Guilfoose JA, Lastinger AM, Smith CL, Arcega VA, Stanley JE, Summerfield HM, Fisher-Duda C, Nepal M, Wen S, Sarwari AR. Using the Comparing Oral versus Parenteral Antimicrobial Therapy (COPAT) Clinical Trial to Influence Institutional Practice Transformation Towards Earlier Transition to Oral Antibiotics. Clin Infect Dis. 2025 Dec 19:ciaf707. doi: 10.1093/cid/ciaf707. Online ahead of print. PMID 41419216
- [Background] Juskowich JJ, Thompson JM, Guilfoose JG, et al. P-106. Preliminary Results of the Comparing Oral versus Parenteral Antimicrobial Therapy (COPAT) Clinical Trial. Open Forum Infect Dis 2025;12(1):S197-198.
- [Background] Juskowich JJ, Thompson JM, Sarwari AR. 333. How the COVID-19 Pandemic Accelerated Development of our Complex Outpatient Oral Antimicrobial Therapy (COpAT) Program. Open Forum Infect Dis 2023;10(2):S212.
- [Background] Juskowich JJ, Ward A, Spigelmyer AE, et al. 1002. Complex Outpatient Antimicrobial Therapy (COpAT) Program at a Rural Academic Medical Center: Evaluation of First 100 Patients. Open Forum Infect Dis 2022;9(2):S418-S419.
- [Background] Kaasch AJ, Lopez-Cortes LE, Rodriguez-Bano J, Cisneros JM, Dolores Navarro M, Fatkenheuer G, Jung N, Rieg S, Lepeule R, Coutte L, Bernard L, Lemaignen A, Kosters K, MacKenzie CR, Soriano A, Hagel S, Fantin B, Lafaurie M, Talarmin JP, Dinh A, Guimard T, Boutoille D, Welte T, Reuter S, Kluytmans J, Martin ML, Forestier E, Stocker H, Vitrat V, Tattevin P, Rommerskirchen A, Noret M, Adams A, Kern WV, Hellmich M, Seifert H; SABATO study group. Efficacy and safety of an early oral switch in low-risk Staphylococcus aureus bloodstream infection (SABATO): an international, open-label, parallel-group, randomised, controlled, non-inferiority trial. Lancet Infect Dis. 2024 May;24(5):523-534. doi: 10.1016/S1473-3099(23)00756-9. Epub 2024 Jan 17. PMID 38244557
- [Background] Kaasch AJ, Barlow G, Edgeworth JD, Fowler VG Jr, Hellmich M, Hopkins S, Kern WV, Llewelyn MJ, Rieg S, Rodriguez-Bano J, Scarborough M, Seifert H, Soriano A, Tilley R, Torok ME, Weiss V, Wilson AP, Thwaites GE; ISAC, INSTINCT, SABG, UKCIRG, and Colleagues. Staphylococcus aureus bloodstream infection: a pooled analysis of five prospective, observational studies. J Infect. 2014 Mar;68(3):242-51. doi: 10.1016/j.jinf.2013.10.015. Epub 2013 Nov 16. PMID 24247070
- [Background] Li HK, Rombach I, Zambellas R, Walker AS, McNally MA, Atkins BL, Lipsky BA, Hughes HC, Bose D, Kumin M, Scarborough C, Matthews PC, Brent AJ, Lomas J, Gundle R, Rogers M, Taylor A, Angus B, Byren I, Berendt AR, Warren S, Fitzgerald FE, Mack DJF, Hopkins S, Folb J, Reynolds HE, Moore E, Marshall J, Jenkins N, Moran CE, Woodhouse AF, Stafford S, Seaton RA, Vallance C, Hemsley CJ, Bisnauthsing K, Sandoe JAT, Aggarwal I, Ellis SC, Bunn DJ, Sutherland RK, Barlow G, Cooper C, Geue C, McMeekin N, Briggs AH, Sendi P, Khatamzas E, Wangrangsimakul T, Wong THN, Barrett LK, Alvand A, Old CF, Bostock J, Paul J, Cooke G, Thwaites GE, Bejon P, Scarborough M; OVIVA Trial Collaborators. Oral versus Intravenous Antibiotics for Bone and Joint Infection. N Engl J Med. 2019 Jan 31;380(5):425-436. doi: 10.1056/NEJMoa1710926. PMID 30699315
- [Background] Comba IY, Go JR, Vaillant J, O'Horo JC, Stevens RW, Palraj R, Abu Saleh O. Sequential Time to Positivity as a Prognostic Indicator in Staphylococcus aureus Bacteremia. Open Forum Infect Dis. 2024 Mar 21;11(4):ofae173. doi: 10.1093/ofid/ofae173. eCollection 2024 Apr. PMID 38617074
- [Background] Cao Y, Guimaraes AO, Peck MC, Mayba O, Ruffin F, Hong K, Carrasco-Triguero M, Fowler VG Jr, Maskarinec SA, Rosenberger CM. Risk stratification biomarkers for Staphylococcus aureus bacteraemia. Clin Transl Immunology. 2020 Feb 13;9(2):e1110. doi: 10.1002/cti2.1110. eCollection 2020. PMID 32082571
- [Background] Bai AD, Lo CKL, Komorowski AS, Suresh M, Guo K, Garg A, Tandon P, Senecal J, Del Corpo O, Stefanova I, Fogarty C, Butler-Laporte G, McDonald EG, Cheng MP, Morris AM, Loeb M, Lee TC. Staphylococcus aureus bacteraemia mortality: a systematic review and meta-analysis. Clin Microbiol Infect. 2022 Aug;28(8):1076-1084. doi: 10.1016/j.cmi.2022.03.015. Epub 2022 Mar 23. PMID 35339678
- [Background] Honda H, Krauss MJ, Jones JC, Olsen MA, Warren DK. The value of infectious diseases consultation in Staphylococcus aureus bacteremia. Am J Med. 2010 Jul;123(7):631-7. doi: 10.1016/j.amjmed.2010.01.015. Epub 2010 May 20. PMID 20493464
- [Background] Iversen K, Ihlemann N, Gill SU, Madsen T, Elming H, Jensen KT, Bruun NE, Hofsten DE, Fursted K, Christensen JJ, Schultz M, Klein CF, Fosboll EL, Rosenvinge F, Schonheyder HC, Kober L, Torp-Pedersen C, Helweg-Larsen J, Tonder N, Moser C, Bundgaard H. Partial Oral versus Intravenous Antibiotic Treatment of Endocarditis. N Engl J Med. 2019 Jan 31;380(5):415-424. doi: 10.1056/NEJMoa1808312. Epub 2018 Aug 28. PMID 30152252
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Background] Liu C, Strnad L, Beekmann SE, Polgreen PM, Chambers HF. Clinical Practice Variation Among Adult Infectious Disease Physicians in the Management of Staphylococcus aureus Bacteremia. Clin Infect Dis. 2019 Jul 18;69(3):530-533. doi: 10.1093/cid/ciy1144. PMID 30601989
- [Background] Minejima E, Mai N, Bui N, Mert M, Mack WJ, She RC, Nieberg P, Spellberg B, Wong-Beringer A. Defining the Breakpoint Duration of Staphylococcus aureus Bacteremia Predictive of Poor Outcomes. Clin Infect Dis. 2020 Feb 3;70(4):566-573. doi: 10.1093/cid/ciz257. PMID 30949675
- [Background] Mourad A, Nwafo N, Skalla L, Holland TL, Jenkins TC. Oral Versus Intravenous Antibiotic Therapy for Staphylococcus aureus Bacteremia or Endocarditis: A Systematic Review and Meta-Analysis of Randomized, Controlled Trials. Clin Infect Dis. 2025 Feb 5;80(1):29-36. doi: 10.1093/cid/ciae476. PMID 39290168
- [Background] Pries-Heje MM, Wiingaard C, Ihlemann N, Gill SU, Bruun NE, Elming H, Povlsen JA, Madsen T, Jensen KT, Fursted K, Schultz M, Ostergaard L, Christensen JJ, Christiansen U, Rosenvinge F, Helweg-Larsen J, Fosbol EL, Kober L, Torp-Pedersen C, Tonder N, Moser C, Iversen K, Bundgaard H. Five-Year Outcomes of the Partial Oral Treatment of Endocarditis (POET) Trial. N Engl J Med. 2022 Feb 10;386(6):601-602. doi: 10.1056/NEJMc2114046. No abstract available. PMID 35139280
- [Background] Swets MC, Bakk Z, Westgeest AC, Berry K, Cooper G, Sim W, Lee RS, Gan TY, Donlon W, Besu A, Heppenstall E, Tysall L, Dewar S, de Boer M, Fowler VG Jr, Dockrell DH, Thwaites GE, Pujol M, Pallares N, Tebe C, Carratala J, Szubert A, Groeneveld GH, Russell CD. Clinical Subphenotypes of Staphylococcus aureus Bacteremia. Clin Infect Dis. 2024 Nov 22;79(5):1153-1161. doi: 10.1093/cid/ciae338. PMID 38916975
- [Background] Percival KM. The Changing Landscape of OPAT to COpAT. Haelio: Infectious Diseases News. May 9, 2023. Accessed May 10, 2023.